CLINICAL TRIAL: NCT01573299
Title: Ischemic Stroke and Early Vertical Positioning, the SEVEL Study: a Randomised Controlled Trial Comparing the 3 Months Rankin Score Outcome in Ischemic Stroke Patients; in Whom Early or Delayed Mobilization is Performed
Brief Title: Ischemic Stroke and Early Vertical Positioning (SEVEL)
Acronym: SEVEL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The required number of patients was not reached. The sites were not able to include more patients.Despite several actions the stop of the study has been decided
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 11/4-C
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Early Mobilisation in Ischemic Stroke Patients
Keywords: Cerebral Infarction, Mobilization, Recovery
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early vertical positioning (Active Comparator)
  Interventions: Other: Mobilization of stroke patients
- Progressively vertical positioning (Active Comparator)
  Interventions: Other: Mobilization of stroke patients

INTERVENTIONS:
Other: Mobilization of stroke patients — In the first group (early vertical positioning)the patient can sit outside of the bed, the day after stroke onset. In the second group (progressively vertical positioning), the patient is progressively "verticalised" and is allowed to sit outside of the bed on the third day after the stroke onset.

SUMMARY:
Even if it is a daily questioning for the stroke physician, no concrete recommendation exists regarding the time-point of the mobilization of stroke patients. In this study, we will compare two mobilisation strategies: early versus delayed "verticalisation". 400 ischemic stroke patients will be included in this prospective randomized controlled trial, equally distributed in two groups. In the early mobilisation procedure the patient is allowed to go and sit outside of the bed the day after the stroke onset, whereas in the other arm, this procedure is delayed to the third day after stroke onset. The outcome in both groups will be assessed by the modified Rankin Scale at 3 months, which is commonly used in stroke study to investigate the functional outcome of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Persistent neurological impairment at the participated time, related to an ischemic stroke defined by a sudden neurological deficit. The neurological deficit must not accompany hemorrhage on cerebral tomodensitometry which occurs on the same day or the day previous to the participation
* Patient hospitalized in Neurology department on the day of the participation
* Patient affiliated to the social security

Exclusion Criteria:

* Malignant cerebral infarction, loss of consciousness, comatose with GCS under 13, cerebral herniation, life- threatening infarction.
* Minor neurological deficit defined by isolated facial palsy, dysarthria, hemianopia, sensitive impairment, or every clinical condition that let the physician thinks that the stay in the hospital would be less than 72 hours.
* Known intracranial stenosis above 50% linked to the current infarction
* History of orthostatic neurological degradation
* Vomiting
* Deep venous thrombosis or suspicion of.
* Patients displaying a loss of autonomy with a Rankin score >3 previous to stroke onset.
* Patient's refusal
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To demonstrate that functional modified Rankin score at 3 months after stroke onset is better with an earlier mobilization protocol (Rankin score) | 3 months

SECONDARY OUTCOMES:
To demonstrate that neurological recovery is better at 7 days with an earlier mobilization protocol (NIHSS score) | 7 days
To demonstrate that neurological recovery is better at 3 months with an earlier mobilization protocol (NIHSS score) | 3 months
To demonstrate that functional modified Rankin score at 7 days after stroke onset is better with an earlier mobilization protocol (Rankin score) | 7 days
To demonstrate that the autonomy is better at 7 days in the early mobilization group (Barthel score) | 7 days
To demonstrate that the autonomy is better at 3 months in the early mobilization group (Barthel score) | 3 months
To demonstrate that an earlier " verticalization " shortens the length of stay in hospital | 7 days
To demonstrate that an earlier " verticalization " allows the patient to go back home sooner | 7 days
To assess the tolerance of an early mobilization | 3 months
To assess the impact of an early mobilization on the post stroke fatigue | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Fanny HERISSON, Doctor, Principal Investigator — Nantes University Hospital
Locations (12):
- France (12):
  - University Hospital, Angers
  - Hospital, Châteaubriand
  - Hospital, La Roche-sur-Yon
  - Hospital, Le Mans
  - Hospital, Lorient
  - University Hospital, Nantes
  - Hospital Cornouaille, Quimper
  - University Hospital, Rennes
  - Hospital Yves LeFoll, Saint-Brieuc
  - Hospital, Saint-Nazaire
  - University Hospital, Tours
  - Hospital Bretagne Atlantique, Vannes

REFERENCES:
- [Derived] Herisson F, Godard S, Volteau C, Le Blanc E, Guillon B, Gaudron M; SEVEL study group. Early Sitting in Ischemic Stroke Patients (SEVEL): A Randomized Controlled Trial. PLoS One. 2016 Mar 29;11(3):e0149466. doi: 10.1371/journal.pone.0149466. eCollection 2016. PMID 27023901